CLINICAL TRIAL: NCT02058186
Title: Effect of Oral Vitamin D Supplement on Atopic Dermatitis; A Clinical Trial With Staphylococcus Aureus Colonization Determination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Srinakharinwirot University (Other)
Responsible Party: Principal Investigator, Montree Udompataikul, Skin Center, Srinakharinwirot University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 218/2555
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, vitamin D supplementation, cathelicidin, Staphylococcus aureus colonization, SCORAD score
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Atopic dermatitis patients: Active (Active Comparator): Atopic dermatitis patients: age 1-18 years old
  Interventions: Drug: oral vitamin D
- Atopic dermatitis patients: Placebo (Placebo Comparator): Atopic dermatitis patients: age 1-18 years old
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral vitamin D
  Arms: Atopic dermatitis patients: Active
Drug: Placebo
  Arms: Atopic dermatitis patients: Placebo

SUMMARY:
Background: Increase in skin colonization of Staphylococcus aureus (S. aureus) in atopic dermatitis patients (AD) resulted from the reduction of cathelicidin production in these patients plays the important role in pathogenesis of this disease. Recently in vivo study has showed that vitamin D can stimulate cathelicidin production. Oral supplement of vitamin D might be beneficial in atopic dermatitis.

Objective: To determine the effect of oral vitamin D supplement on clinical impact including skin colonization of S. aureus in atopic dermatitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Eligible criteria included patients with mild to moderate atopic dermatitis by SCORAD (Scoring for Atopic Dermatitis) score criteria1,17,18, age between 1-18 years old. All patients had been advised to take normal, dietary product and their activities. They had been advised to discontinue at least 4 weeks of oral corticosteroid, at least 2 weeks of topical corticosteroid or topical calcineurin inhibitor application and at least 6 months of vitamin supplement prior to starting the protocol

Exclusion Criteria:

* The exclusion criteria were to coexisting skin infection on top with AD lesions, known case of primary or secondary immune-compromised host, hepatic or renal disease, those taking vitamin D or nutraceutical supplementation, those continues taking with antibiotics, corticosteroid, immunosuppressive agents, anti-epileptic drugs, thiazide diuretics, proton-pump inhibitors, histamine 2-receptor antagonists at the time of enrollment. Patients who used topical antiseptic or antibiotic products during study period were also excluded. Patients who developed worsening of AD with flare-up of clinical manifestation or SCORAD greater than 40, secondary infection on-top tested lesions were excluded from data analysis.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
SCORAD score | May - August 2012 (3 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Center, Srinakharinwirot University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842